CLINICAL TRIAL: NCT01362465
Title: Characterization of Interventricular Conduction Measurements
Acronym: ICM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TDSICM
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Resynchronization Therapy (CRT) (Experimental): Implanting device to measure delays between paced chambers in heart failure patients.
  Interventions: Procedure: Cardiac Resynchronization Therapy

INTERVENTIONS:
Procedure: Cardiac Resynchronization Therapy — Implanting device to measure delays between paced chambers in heart failure patients.
  Other Names: CRT

SUMMARY:
This study is an effort to use left ventricular (LV) lead based measurements to identify late electrical activation and avoid scar.

DETAILED DESCRIPTION:
The aim of this study is to characterize how right ventricular (RV) to left ventricular (LV) conduction delays are altered by pacing site in patients with a cardiac resynchronization therapy (CRT) system. The study will be performed in conjunction with a CRT implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than 18 years of age.
* The patient or the patient's legally authorized representative is willing to give informed consent.
* CRT indicated guidelines.
* Patient is receiving a Medtronic IPG or ICD.

Exclusion Criteria:

* Patients who are pregnant.
* Patient is in AF.
* Patient with 3rd degree AV block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measure how RV to LV conduction times are altered by pacing site in patients with a CRT system. | 30 minutes
  This procedure will take approximately 30 minutes prior to implant of a CRT system. At completion of this study the patient is not followed and will be transferred to another study if enrolled in a clinical or followed as a routine implant by the center.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Atwater, MD, Principal Investigator — Durham VA; Robert Hoyt, MD, Principal Investigator — Catholic Health Initiative Iowa Corp; Eric E Johnson, MD, Principal Investigator — Sterns Cardiovascular Foundation; John F Beshai, MD, Principal Investigator — University of Chicago